CLINICAL TRIAL: NCT06475846
Title: A Evaluate HRS5580 for Injection for Prevention of Postoperative Nausea and Vomiting Efficacy and Safety of Ⅱ Period, Randomized, Multicenter, Dose of Exploration, Positive Control, Placebo-controlled, Double-blind, Double Simulation Trials
Brief Title: A Trial of HRS5580 in Prevention of Postoperative Nausea and Vomiting of Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Shengdi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS5580-201
Record Dates: First submitted 2024-06-13; First posted 2024-06-26 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Preventing of Postoperative Nausea and Vomiting in Adults
MeSH Terms: interventions — Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Treatment group A: HRS5580 (Experimental)
  Interventions: Drug: HRS5580
- Treatment group B: HRS5580 (Experimental)
  Interventions: Drug: HRS5580
- Treatment group C: HRS5580 (Experimental)
  Interventions: Drug: HRS5580
- Treatment group D: Ondansetron (Active Comparator)
  Interventions: Drug: Ondansetron
- Treatment group E: blank preparation. (Placebo Comparator)
  Interventions: Drug: blank preparation

INTERVENTIONS:
Drug: HRS5580 — HRS5580; low dose
  Arms: Treatment group A: HRS5580
Drug: HRS5580 — HRS5580; middle dose
  Arms: Treatment group B: HRS5580
Drug: HRS5580 — HRS5580; middle dose
  Arms: Treatment group C: HRS5580
Drug: Ondansetron — Ondansetron
  Arms: Treatment group D: Ondansetron
Drug: blank preparation — blank preparation.
  Arms: Treatment group E: blank preparation.

SUMMARY:
The study is being conducted to evaluate the efficacy, and safety of HRS5580 for preventing of postoperative nausea and vomiting in adults. To explore the reasonable dosage of HRS5580 for postoperative nausea and vomiting.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent
2. Plan to undergo elective surgery under general anesthesia；
3. ≥18 years old
4. Meet the weight standard
5. Conform to the ASA Physical Status Classification
6. Expected postoperative hospital stay ≥72 hours
7. PONV risk factors ≥3

Exclusion Criteria:

1. Subjects with vomiting and/or retching and nausea occurred before surgery
2. Subjects with a history of vestibular disease, central nervous system and other system diseases
3. Subjects with a previous history of chronic nausea or vomiting/retching
4. Subjects with a history of myocardial infarction or unstable angina pectoris
5. Subjects with atrioventricular block or cardiac insufficiency
6. Subjects with a history of ischemic stroke or transient ischemic attack
7. Subjects with poor blood pressure control after medication
8. Abnormal electrocardiogram
9. Abnormal values in the laboratory
10. Allergic to a drug ingredient or component
11. Received treatment with potential antiemetic effects before starting the investigational product
12. Subjects who received chemotherapy prior to surgery
13. Use of drugs that affect the antiemetic effect, and the time between the last use of the test drug and the start of the time is less than 5 half-lives
14. Plan to receive local anesthesia only or total intravenous anesthesia only
15. Subjects who are expected to require an in-situ nasogastric tube or orogastric tube after completion of surgery
16. Subjects expected to be transferred to the ICU at the end of surgery
17. Pregnant or nursing women
18. No birth control during the specified period of time
19. Participated in clinical trials of other drugs (received experimental drugs)
20. The inestigators determined that other conditions were inappropriate for participation in this clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2024-06-25 (Actual); Primary Completion 2024-10-29 (Actual); Study Completion 2024-10-29 (Actual)

PRIMARY OUTCOMES:
No vomiting rate within 72 hours after extubation | at 72 hours after extubation

SECONDARY OUTCOMES:
Complete response rate (defined as the proportion of subjects without vomiting and receiving no rescue therapy) at 24, 48, 72, 96, and 120 hours after extubation | at24, 48, 72, 96, and 120 hours after extubation
No vomiting at 24, 48, 96, and 120 hours after extubation, | at 24, 48, 96, and 120 hours after extubation
Proportion of subjects who did not experience significant nausea within 24, 48, 72, 96, and 120 hours after extubation | at 24, 48, 72, 96, and 120 hours after extubation
Proportion of participants not receiving rescue medication within 24, 48, 72, 96, and 120 hours of extubation | at 24, 48, 72, 96, and 120 hours of extubation

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Third Xiangya Hospital of Central South University, Changsha, Hu'nan

IPD SHARING:
Plan to Share IPD: Undecided